CLINICAL TRIAL: NCT04702984
Title: Clinical Characterization of an Investigational Frequent Replacement Daily Wear Silicone Hydrogel Sphere Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL949-E003
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Results first posted 2022-03-08 (Actual); Last update posted 2022-03-16 (Actual); Status verified 2022-03

CONDITIONS: Refractive Errors
Keywords: Vision; Contact lenses
MeSH Terms: conditions — Refractive Errors

STUDY DESIGN:
Masking Description: Lens will be provided with investigational product labeling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- LID021201 (Experimental): LID021201 contact lenses worn in both eyes for 7 days. Lenses will be removed nightly for cleaning and disinfection with OPTI-FREE multipurpose solution.
  Interventions: Device: LID021201 contact lenses; Device: OPTI-FREE multipurpose solution

INTERVENTIONS:
Device: LID021201 contact lenses — Investigational silicone hydrogel sphere contact lenses for frequent replacement daily wear
Device: OPTI-FREE multipurpose solution — Solution for cleaning, disinfecting, and reconditioning silicone hydrogel contact lenses
  Other Names: OPTI-FREE® RepleniSH®

SUMMARY:
The primary objective of this study is to evaluate the overall clinical performance of an investigational silicone hydrogel contact lens over 7 days of daily wear.

DETAILED DESCRIPTION:
Participants will attend a Screening visit, a Dispense visit, and a Week 1 Follow-up/exit visit.

ELIGIBILITY:
Inclusion Criteria:

* Understand and sign an Informed Consent that has been approved by an Institutional Review Board.
* Successful wear of spherical daily wear frequent replacement soft contact lenses in both eyes for a minimum of 5 days per week and 8 hours per day during the past 3 months.
* Willing to stop wearing habitual contact lenses for the duration of study participation.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Any condition that contraindicates contact lens wear, as determined by the Investigator.
* Any use of systemic or ocular medications that contraindicates contact lens wear, as determined by the Investigator.
* History of refractive surgery or plan to have refractive surgery during the study.
* Current or history of dry eye in either eye that, in the opinion of the Investigator, would preclude contact lens wear.
* Wears habitual contact lenses in an extended wear modality (routinely sleeping in lenses for at least 1 night per week) over the last 3 months prior to enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2021-01-21 (Actual); Primary Completion 2021-02-26 (Actual); Study Completion 2021-02-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sr. Clinical Trial Lead, CDMA Vision Care, Study Director — Alcon Research, LLC
Locations (3):
- United States (3):
  - Alcon Investigator 6565, Maitland, Florida
  - Alcon Investigator 6353, Memphis, Tennessee
  - Alcon Investigator 8028, Wichita Falls, Texas

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at 3 investigative sites located in the United States.
Pre-assignment Details: This reporting group includes all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used with the purpose of power optimization (Safety Analysis Set).
Units Other Than Participants: eyes
Groups:
- LID021201: LID021201 contact lenses worn in both eyes for 7 days. Lenses were removed nightly for cleaning and disinfection with OPTI-FREE multipurpose solution.
Period: Overall Study
Arm/Group | LID021201
Started | 39; 78 eyes
Completed | 38; 76 eyes
Not Completed | 1; 2 eyes
Not completed — Adverse Event Unrelated to the Study Device | 1

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set
Arm/Group | LID021201
Number analyzed (Participants) | 39
Age, Continuous [Mean (Standard Deviation); unit: years] | 35.1 (7.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Front Surface Wettability, by Category
Description: Front surface wettability (i.e., assessment of the disruption of the front surface wettability of the contact lens) was assessed by the investigator for each eye individually. Front surface wettability was collected on a 5-point scale, where where Grade 0 = a smooth uniformly reflecting surface, Grade 1 = a coarse hazy surface which seems resolved momentarily with each blink and becomes exacerbated with staring, Grade 2 = one stable dry (non-wetting) area of some magnitude, Grade 3 = more than one stable dry (non-wetting) area of some magnitude, and Grade 4 = non-wettable lens surface. No formal hypothesis was predefined for the primary endpoint. No inferential testing was performed.
Time Frame: Dispense; Week 1 Follow-up
Population: Safety Analysis Set
Measure: Number; unit: eyes
Units Other Than Participants: eyes
Arm/Group | LID021201
Number analyzed (Participants) | 39
Number analyzed (eyes) | 78
eyes
  Dispense, Grade 0 | 78
  Dispense, Grade 1 | 0
  Dispense, Grade 2 | 0
  Dispense, Grade 3 | 0
  Dispense, Grade 4 | 0
  Week 1 Follow-up, Grade 0: number analyzed (Participants) | 38
  Week 1 Follow-up, Grade 0: number analyzed (eyes) | 76
  Week 1 Follow-up, Grade 0 | 56
  Week 1 Follow-up, Grade 1: number analyzed (Participants) | 38
  Week 1 Follow-up, Grade 1: number analyzed (eyes) | 76
  Week 1 Follow-up, Grade 1 | 19
  Week 1 Follow-up, Grade 2: number analyzed (Participants) | 38
  Week 1 Follow-up, Grade 2: number analyzed (eyes) | 76
  Week 1 Follow-up, Grade 2 | 1
  Week 1 Follow-up, Grade 3: number analyzed (Participants) | 38
  Week 1 Follow-up, Grade 3: number analyzed (eyes) | 76
  Week 1 Follow-up, Grade 3 | 0
  Week 1 Follow-up, Grade 4: number analyzed (Participants) | 38
  Week 1 Follow-up, Grade 4: number analyzed (eyes) | 76
  Week 1 Follow-up, Grade 4 | 0

ADVERSE EVENTS:
Time Frame: Adverse events (AE's) were collected from time of consent to study exit, approximately 1 week.
Description: AE's were obtained through solicited and spontaneous comments from subjects and through observations by the Investigator. "At Risk" population for ocular AEs is reported in units of eyes; all other populations are reported in units of participants. This analysis population includes all subjects/eyes exposed to any study lenses evaluated in this study, except for the lenses used with the purpose of power optimization.
Groups:
- Pretreatment: Events reported in this group occurred prior to exposure to the study contact lenses
- LID021201 Ocular; LID021201 Nonocular: Events reported in this group occurred while exposed to the study contact lenses
Arm/Group | Pretreatment | LID021201 Ocular | LID021201 Nonocular
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/78 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/78 | 0/39
Other Adverse Events (participants affected / at risk) | 0/39 | 0/78 | 0/39

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.

DOCUMENTS (2):
  • Study Protocol (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/84/NCT04702984/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-13): https://cdn.clinicaltrials.gov/large-docs/84/NCT04702984/SAP_001.pdf